CLINICAL TRIAL: NCT06956768
Title: Helmet Therapy for Positional Cranial Deformities: Any Impact on Skull's Growth?
Brief Title: Head Circumference Evolution in Children With Positional Plagiocephaly During and After Molding Helmet Therapy.
Acronym: PCPlagio
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, STELLA Irène, Neurosurgeon, Central Hospital, Nancy, France
Other Study IDs: CHRU Nancy : 2025PI044
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-03

CONDITIONS: Non Synostotic Plagiocephaly
Keywords: deformational plagiocephaly; cranial circumpherence
MeSH Terms: conditions — Plagiocephaly, Nonsynostotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to verify the growth of cranial circumference in children treated with helmets for positional skull deformity. The main questions it aims to answer are as follows:

Does the helmet produce a reduction in cranial growth during the period in which it is worn? If the growth of the cranial circumference slows down while the helmet is being worn, does it recover a few months after the end of the treatment? The researchers will study changes in cranial circumference during and after helmet treatment.

The participants received helmet treatment as part of their usual medical care. They will be followed until medical attention is required and data will be collected retrospectively.

DETAILED DESCRIPTION:
Cranial positional deformities in children are a major health problem in France, as in other countries, with a reported incidence of up to 47%. This phenomenon started to widespread in the 90s, but widely diffused in France after 2020, following paediatric recommendations for infants to be placed strictly on their backs in order to avoid sudden infant death syndrome.

Cranial deformation may be asymmetrical (plagiocephaly) or symmetrical (brachycephaly), depending on whether or not a torticollis or a positional preference coexist. The consequences of these deformations are mostly aesthetics, giving the fact that there is no brain compression nor sufferance. In some severe cases, compensational skull growth in the temporo-parietal region, uni- or bilaterally, is noticed immediately on frontal face view, accounting for a disgraceful facial appearance. This aspect is source of parental anxiety and distress, with feeling of guilty and fear for the future of their child.

A part from aesthetic consequences, while in brachycephaly, the symmetrical morphology of the skull justifies the fact that there are no functional consequences, in severe plagiocephaly, a skull base displacement may also be observed, with impact on the frontal region and advancement of the ipsilateral frontal bone, and consequent asymmetrical development of the mandibular and cervical musculoskeletal component.

Intensive stimulation of the child, often with the help of physiotherapists, became essential in order to prevent any deformities.

Despite educational efforts and preventive measures, many cases of positional skull deformity still occur and come to the attention of paediatric neurosurgeons. One of the solutions proposed in the most severe cases is the fitting of a custom-made cranial orthosis (helmet), capable to guide the remodelling of the skull and to reduce the deformity. As with all medical devices, the cranial orthosis is not without its risks and complications. Some of these complications, such as frontal skin burnt at helmet compression points, have already been widely described in the literature.

From personal experience, in patients who have been monitored while wearing the orthosis, it has been frequently observed an inflection of the curve of the cranial perimeter (CP) corresponding to the time the helmet is worn. For this reason, it is essential to measure the CP curve in children who have benefited from a helmet, in order to check that growth has restored some months after the treatment. Anyway, even if CP's reduction is minimal and spontaneously corrects, it is necessary for health care professionals and orthoprosthetist to be aware of this phenomenon, which implies a certain degree of cranial compression during helmet therapy.

ELIGIBILITY:
Inclusion Criteria:

* Children under 12 months of age with diagnosis of positional deformity of the cranium.
* Treated with a cranial orthosis.

Exclusion Criteria:

* Children with orthoses fitted before the consultation.
* Children whose parents have not authorised data analysis.

Ages: 4 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Referred to the Craniost Reference Center for Rares Diseases of the Nancy Regional University Hospital for a positional deformity of the cranium.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Cranial circumpherence curve | 6 months after the the end of the treatment.
  Evaluation of changes in standard deviations of head circumference during and after wearing the helmet.
  Measurement of cranial perimeter (CP):
  * Value expressed in cm.
  * Traceable on a standardised record curve; each value corresponds to a precise standard deviation (SD) on the curve: - 2SD, - 1.5SD, - 1SD, -0.5 SD, 0SD, + 0.5 SD, + 1SD, + 1.5SD, + 2SD.

SECONDARY OUTCOMES:
Complications | From the beginning to 6 months after the the end of the treatment.
  Note the presence of any other complications that arose while wearing the helmet (yes/no):
  * Skin burns;
  * Slower acquisition;
  * Intolerance;
  * Other.
Morphological aspects | From the enrollement to 6 months after the the end of the treatment.
  Evaluate the changes in the cranial indexes after treatment with the orthosis.
  * Cranial Index (CI) = biparietal cranial diameter (LL)/ antero-posterior cranial diameter (AP)
  * Cranial Vault Asymetry Index (CVAI) = major cranial diagonal (D1) - minor cranial diagonal (D2) x 100/D1
  Values are expressed in cm.
Aesthetics features | From the enrollement to 6 months after the end of the treatment
  Assess the presence of morphological severity criteria (yes/no): ear asymmetry, frontal asymmetry, compensatory growth.
Radiological features | 6 months after the the end of the treatment.
  Evaluation of CT scans: presence of ptosis of the cerebellar tonsils (yes/no); presence of asymmetry of the base of the skull (yes/no).
Radiological features | From the enrollement to 6 months after the end of the treatment
  Measurement of posterior fossa volume

IPD SHARING:
Plan to Share IPD: Undecided
I would like to share for transparency policy, but I don't have discussed yet with our data commitee.

REFERENCES:
- [Background] Ballardini E, Sisti M, Basaglia N, Benedetto M, Baldan A, Borgna-Pignatti C, Garani G. Prevalence and characteristics of positional plagiocephaly in healthy full-term infants at 8-12 weeks of life. Eur J Pediatr. 2018 Oct;177(10):1547-1554. doi: 10.1007/s00431-018-3212-0. Epub 2018 Jul 20. PMID 30030600
- [Background] Picart T, Beuriat PA, Szathmari A, Di Rocco F, Mottolese C. Positional cranial deformation in children: A plea for the efficacy of the cranial helmet in children. Neurochirurgie. 2020 Apr;66(2):102-109. doi: 10.1016/j.neuchi.2019.10.011. Epub 2020 Jan 17. PMID 31958410
- [Background] Kreutz M, Fitze B, Blecher C, Marcello A, Simon R, Cremer R, Zeilhofer HF, Kunz C, Mayr J. Facial asymmetry correction with moulded helmet therapy in infants with deformational skull base plagiocephaly. J Craniomaxillofac Surg. 2018 Jan;46(1):28-34. doi: 10.1016/j.jcms.2017.10.013. Epub 2017 Oct 16. PMID 29221913
- See also: Official High Health Authority of France document. — https://www.has-sante.fr/jcms/p_3151574/fr/prevention-des-deformations-craniennes-positionnelles-dcp-et-mort-inattendue-du-nourrisson